CLINICAL TRIAL: NCT04933110
Title: Investigation of Hand Functions and Related Parameters in People With Multiple Sclerosis in the Very Early Stage.
Brief Title: Investigation of Hand Functions and Related Parameters in People With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uğur OVACIK (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor-Investigator, Uğur OVACIK, Principal Investigator, PT, Msc, Istanbul Aydın University
Organization: Istanbul Aydın University (Other)
Other Study IDs: İAÜ2
Record Dates: First submitted 2021-06-14; First posted 2021-06-21 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; upper limb function; activity; participation
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis: Individuals with early-stage multiple sclerosis
- Healthy Volunteers: Healthy volunteers of similar age and sex as individuals with multiple sclerosis

SUMMARY:
The upper extremity in people with Multiple Sclerosis (pwMS) has become a more popular research topic in recent years, with the increase in studies reporting widespread involvement. The aim of our study was to evaluate the upper extremity from multiple perspectives in early stage pwMS, to identify problems by comparing them with healthy individuals, and to examine the relationship of problems with activity and participation.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis according to McDonald criteria
* Relapsing Remitting MS clinical course type
* 18-65 age range
* Being able to understand and read Turkish

Exclusion Criteria:

* Having an MS attack in the last 3 months
* To have done regular exercise for the upper extremity in the 6 months before starting the study
* Having different neurological, orthopedic or cardiac problems other than MS
* Being addicted to alcohol or drugs
* Getting a score below 24 on the Mini Mental Test Scale
* Having a spasticity of 3 or more according to the Modified Ashworth Scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with MS who met the inclusion criteria and volunteered to participate in the study.
  Volunteer healthy individuals of similar age and sex with individuals with MS.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-07-05 (Estimated); Primary Completion 2021-09-06 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Nine Hole Peg Test | baseline (on the predetermined assessment day)
  To assess upper extremity function. Completing the test in a short time (seconds) indicates better upper extremity function.
Minnesota Manual Dexterity Test | baseline (on the predetermined assessment day)
  To assess upper extremity function. Completing the test in a short time (seconds) indicates better upper extremity function.
ABILHAND | baseline (on the predetermined assessment day)
  To assess for performance of activity. Score range 0-46 point, higher scores mean a better outcome.
Motor Activity Log-28 | baseline (on the predetermined assessment day)
  To assess for performance of activity. Score range 0-5 point, a high score indicates good upper extremity use frequency and quality of movement during activity.
Community Integration Questionnaire | baseline (on the predetermined assessment day)
  To assess participation. The total score ranges from 0-29, and the higher the score, the higher the individual's participation in society is considered.

SECONDARY OUTCOMES:
Hand Held Dynamometer | baseline (on the predetermined assessment day)
  To assess upper extremity muscle strength. Higher scores indicate better muscle strength.
Hand Dynamometer | baseline (on the predetermined assessment day)
  To assess grip strength. Higher scores indicate better muscle strength.
Pinchmeter | baseline (on the predetermined assessment day)
  To assess pinch strength. Higher scores indicate better muscle strength.
Tuning fork | baseline (on the predetermined assessment day)
  To assess deep sense. A higher score indicates better sensitivity.
Aesthesiometer | baseline (on the predetermined assessment day)
  To assess two-point discrimination. A higher score indicates worse sensitivity.
Fatigue Severity Scale | baseline (on the predetermined assessment day)
  To assess the severity of fatigue. Score range 1-7 point, a higher score indicates more severe fatigue.
Symbol Digit Modalities Test | baseline (on the predetermined assessment day)
  To assess cognitive level. A higher score indicates better cognitive level.
Hospital Anxiety and Depression Scale | baseline (on the predetermined assessment day)
  To assess anxiety and depression. The total score ranges from 0 to 21 for each of the two subscales. A higher score indicates more severe anxiety and depression.